CLINICAL TRIAL: NCT05894772
Title: Evaluating a Virtual Stepped Care Portal in Youth Awaiting Tertiary Chronic Pain Care: An Implementation-Effectiveness Hybrid Type III Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Calgary (Other); University of Saskatchewan (Other); Centre for Addiction and Mental Health (Other); University of British Columbia (Other); Memorial University of Newfoundland (Other); University of Alberta (Other); St. Justine's Hospital (Other); McMaster Children's Hospital (Other); Dalhousie University (Other); Montreal Children's Hospital of the MUHC (Other); Children's Hospital of Eastern Ontario (Other); Provincial Health Services Authority British Columbia (Other); Seattle Children's Hospital (Other); University Health Network, Toronto (Other); London Health Sciences Centre (Other); Quebec Pain Research Network (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Senior Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4025
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Implementation-effectiveness quasi-experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Power over Pain Portal
  Interventions: Behavioral: Power over Pain Portal

INTERVENTIONS:
Behavioral: Power over Pain Portal — Youth from different ages, sexes, gender, sexual orientations, races, dwelling and school/employment status will receive access to the Power over Pain Portal for 4 months. The portal consists of self-assessment tools (bi-weekly check-ins to provide users with feedback on their mood, anxiety, pain, and sleep and guide decision making on choice of interventions), evidence-based virtual educational (pain neuroscience) and cognitive behavioural therapy (CBT) pain interventions that are delivered in a stepped care manner based on participant needs/preference. The overall objective is to determine the implementation (guided by Proctor's implementation conceptual framework) and clinical effectiveness of the PoP Portal in a sample of youth (12-18 years of age) who are on the waitlist for tertiary care consultation at any pediatric CP clinic in Canada.

SUMMARY:
Pain is one of the most common symptoms of extreme stress in youth. Without treatment, short-term pain can last for months to years (called 'chronic pain'; CP), a problem already affecting 1 in 5 Canadian youth. The COVID-19 pandemic is one of the greatest threats to youth mental health seen in generations. CP in childhood can trigger a wave of mental health issues that last well into adulthood. In 2019, we learned that "access to pain care" is poor and a priority for youth with CP and their families. Unfortunately, COVID-19 has only made access more difficult. In 2020, we created an online "stepped care" program called the Power over Pain Portal for youth with CP. Stepped care is a promising way to improve access to CP care by tailoring care based on the symptoms each youth is experiencing. Like a ladder, youth start with one type of care and then "step up" or "step down" to more or less intense care depending on what they need. Over the past year, funded by CIHR, we worked with hundreds of youth and healthcare professionals across Canada to understand how the pandemic has affected pain and mental health. We also summarized all online pain self-management programs including peer support for youth to find the best resources to include in the Portal and will translate the portal content into French. Together with a diverse group of youth with CP, we have now co-designed the online Portal. The next step (focus of this grant) is to test the Portal with youth to ensure it can be implemented and is helpful. We will recruit 93 youth with CP waiting for specialist care at 11 CP clinics across Canada to use the Portal for 4 months. We will see how they use the Portal and if it helps to improve their pain and mental health. This study is important because it will allow us to understand how the Portal works in the real world before wide public release (English and French) to support all youth in Canada with CP with accessible, evidence-based pain care.

ELIGIBILITY:
Inclusion Criteria:

* Experience chronic pain
* Speak and read English or French
* Have access to internet / smartphone (or are willing to be loaned a study phone with a data plan)
* Are on the waitlist of a tertiary care CP clinic in Canada
* Intend to use the PoP Portal for at least 4 months
* Have the capacity to consent

Exclusion Criteria:

* Have moderate to severe cognitive impairments that may impact their ability to understand and use the PoP Portal or complete self-reported clinical outcome measures
* Have untreated major psychiatric illness (e.g., anorexia, psychosis) and/or active suicidality as assessed by the PoP Portal screening. Youth who have co-occurring clinically significant anxiety or depression that is currently being treated will be eligible if they meet other inclusion criteria.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 16 weeks
  Will be assessed using the Acceptability e-Scale administered at T2 and during the qualitative interview. Participants rate features of the portal on a scale from 1-5 with higher scores indicating higher acceptability.
Adoption | 16 weeks
  Characterized via participant-level analytics of interactions with each feature. The benchmark will be >60% of participants completing ≥ 1 portal intervention.
Appropriateness | 16 weeks
  Perceived fit and compatibility of portal participants' needs. Assessed via the qualitative interview at T2.
Portal Feasibility | 16 weeks
  Degree to which to PoP Portal could be used as intended. Will be assessed via monthly audit of support tickets and characterization of the severity of encountered issues.
Fidelity | 16 weeks
  Degree to which the PoP Portal and each intervention independently (WEBMap, iCanCope, iPeer2Peer) was used as intended. Will be characterized by intervention use analytics.

SECONDARY OUTCOMES:
Pain Intensity | 16 weeks
  Will be measured using the PROMIS Pain Intensity Scale which assesses pain the past 7 days using an 11-point numerical rating scale (NRS) with verbal anchors "no pain" at 0 and "worst pain you can think of" at 10. This tool demonstrates relevance, feasibility, and understandability for youth with chronic pain.
Pain Interference | 16 weeks
  Will be assessed using the PROMIS Pain Interference Short-form Scale and 8-item tool that uses a 5-point Likert scale, ranging from never to almost always, with higher scores representing greater interference with function.
Anxiety | 16 weeks
  Will be assessed using a PROMIS Paediatric Anxiety Short-form Scale, an 8-item tool that uses a 5-point Likert scale, ranging from never to almost always, with higher scores representing more anxiety symptoms.
Depression | 16 weeks
  Will be assessed using PROMIS Paediatric Depression Short-form Scale, an 8-item tool that used a 5-point Likert scale, ranging from never to almost always, with higher scores representing more depressive symptoms.
Insomnia | 16 weeks
  Will be assessed using a 7-item Insomnia Severity Index, higher score representing more severe insomnia.
Health Related Quality of Life | 16 weeks
  Will be assessed using a 7-item PROMIS Paediatric Global Health Short-form Scales with higher scores representing overall better health.
School Attendance | 16 weeks
  Will be assessed using a single item modified by investigators to capture school absenteeism as a continuous variable ranging from 0 to 240 days. Self-report of school attendance among a CP population is comparable to school administrative data.
Healthcare Utilization | 16 weeks
  Will capture family physician and emergency visits, psychological or physical therapies and changes in medication, using a CP modified version of Ambulatory and Home Care Record at T1 and T2.

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (11):
  - IWK Health Center, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital London Health Sciences, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Jim Pattison, Saskatoon, Saskatchewan
  - Alberta Children's Hospital, Calgary
  - Stollery Children's Hospital, Edmonton
  - Montreal Children's Hospital, Montreal
  - BC Children's Hospital, Vancouver